CLINICAL TRIAL: NCT03962569
Title: Early Activation of Artificial Urinary Sphincter: A Pilot Study
Brief Title: Early Activation of Artificial Urinary Sphincter
Acronym: WV_AUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Joshua Lohri, Principal Investigator, CAMC Health System
Other Study IDs: 19-556
Record Dates: First submitted 2019-05-17; First posted 2019-05-24 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Incontinence, Urinary
Keywords: Artificial Urinary Sphincter
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary incontinence or loss of bladder control is a troublesome issue for all affected patients. The causes of urinary incontinence and its treatment options vary widely. A commonly encountered reason for urinary incontinence in men is related to treatment for prostate cancer. These treatment options can range from surgical removal of the prostate, external beam radiation therapy, and/or brachytherapy, the insertion of radioactive implants directly into the tissue. Mild cases of incontinence are responsive to more conservative measures, but moderate to severe cases often require placement of an artificial urinary sphincter. Typically, these devices are left deactivated for a period of 4- 6 weeks following implantation to allow swelling to subside before use. The investigators hypothesize that the device could be activated within an earlier timeframe without increasing the risk of complications. No studies to date have evaluated this; therefore the investigators plan to conduct a prospective study in which the investigators will activate the device 3 weeks after placement and monitor for complications.

DETAILED DESCRIPTION:
This study is a single institute prospective study with patients undergoing artificial urinary sphincter placement by the operating surgeon, Dr. Joshua Lohri at Charleston Area Medical Center in Charleston, WV. Any male patients with moderate to severe urinary incontinence who have been treated for prostate cancer (radical prostatectomy, External Beam Radiation therapy or brachytherapy, or Incontinence related to trans urethral resection of the prostate (TURP) or simple prostatectomy undergoing artificial urinary sphincter placement at Charleston Area Medical Center by Dr. Joshua Lohri, D.O. will be offered the chance to participate in this study. The investigators aim to enroll 25 patients, which is anticipate to be accrued within 3 years from the start of the study. Patients will be excluded if: 1) the have previously undergone artificial urinary sphincter placement and presents for revision or additional cuff placement, 2) has had combined artificial urinary sphincter and inflatable penile prosthesis placemen and 3) are a poor candidate for early activation due to poor condition at presentation or signs of infection.

All patients agreeing to participate will have the urinary sphincter activated 3 weeks after surgery. If there are patients that later choose not to have early activation or are found to be poor candidates for three week activation based upon post op exam, the investigator will proceed with activation at a 4-6 week time period. While there is no comparison group in the study, patient satisfaction and adverse events for study patients will be compared to historical literature.

Before the procedure is performed all eligible patients will be informed about the study at the regularly scheduled pre-operative office visit and if the patient would like to participate will be offered to sign the consent document. The participant will receive a copy of the signed consent form and be asked to an SF-8 quality of life survey and Incontinence Impact Questionnaire. Once consented, the patient will undergo the procedure without any changes to the normal routine. The patient's device will be deactivated at the conclusion of the procedure.

After the procedure, the patient will be discharged post-operatively (same day) and follow-up will be arranged in 3 weeks to activate the device (up to 3 weeks and 3 days after the procedure) which includes a post-operative evaluation of incisions, degree of bruising, tissue induration, tenderness and accessibility of the pump. If these factors are acceptable and pump mechanics are normal, the artificial sphincter will be activated and the patient will be educated on its proper use. Additional follow up will include the regular 6 week visit, a visit at 3 months, and then every 6 months for a total of 1 year unless issues arise that necessitates deviation. At each visit, patients will complete the Incontinence Impact Questionnaire and the SF-8 quality of life survey.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing artificial urinary sphincter (AUS) placement by single surgeon, Joshua Lohri, DO.

Exclusion Criteria:

* Any patient who has previously undergone artificial urinary sphincter placement and presents for revision or additional cuff placement.
* Any patient who is undergoing combined artificial urinary sphincter and inflatable penile prosthesis placement.
* Any patient who is a poor candidate for early activation due to poor condition at presentation or signs of infection.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with moderate to severe urinary incontinence
Study Population: All male patients with moderate to severe urinary incontinence who have been treated for prostate cancer (radical prostatectomy, External Beam Radiation therapy or brachytherapy, or Incontinence related to trans urethral resection of the prostate (TURP) or simple prostatectomy undergoing artificial urinary sphincter placement at Charleston Area Medical Center by Dr. Joshua Lohri, D.O.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Incontinence Questionnaire Short form IIQ-7 | pre-procedure, 3 week, 6 week, 3 month, 6 month, 1 year
  patients with earlier AUS activation will have percentage of interference changed scores on the Urinary incontinence survey beginning at 6 week mark and increasing there after until 1 year. Survey includes 7 questions with results values ranging from '0' for no interference up to '3' for greatly interfering in the patient's activities, relationships, and feelings. Higher percentage scores indicate more interference in these activities.
Improved quality of life scores (SF8 4 Week version) | pre-procedure, 3 week, 6 week, 3 month, 6 month, and 1 year
  patients with earlier AUS activation will have changed SF8 scores beginning at 6 week mark and increasing there after due to early activation. Higher scores indicate better self reported quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: joshua lohri, DO, Principal Investigator — CAMC Health System
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Must get approval from CAMC Privacy Office prior to sharing

REFERENCES:
- [Background] Wolin KY, Luly J, Sutcliffe S, Andriole GL, Kibel AS. Risk of urinary incontinence following prostatectomy: the role of physical activity and obesity. J Urol. 2010 Feb;183(2):629-33. doi: 10.1016/j.juro.2009.09.082. Epub 2009 Dec 16. PMID 20018324
- [Background] Viers BR, Linder BJ, Rivera ME, Rangel LJ, Ziegelmann MJ, Elliott DS. Long-Term Quality of Life and Functional Outcomes among Primary and Secondary Artificial Urinary Sphincter Implantations in Men with Stress Urinary Incontinence. J Urol. 2016 Sep;196(3):838-43. doi: 10.1016/j.juro.2016.03.076. Epub 2016 Mar 17. PMID 26997310
- [Background] Parrillo, Lisa.;Wein, Alan. Post Prostatecomy Incontinence. Prostate Cancer (Second Edition), 2016
- [Background] Linder BJ, Piotrowski JT, Ziegelmann MJ, Rivera ME, Rangel LJ, Elliott DS. Perioperative Complications following Artificial Urinary Sphincter Placement. J Urol. 2015 Sep;194(3):716-20. doi: 10.1016/j.juro.2015.02.2945. Epub 2015 Mar 14. PMID 25776908
- [Background] James MH, McCammon KA. Artificial urinary sphincter for post-prostatectomy incontinence: a review. Int J Urol. 2014 Jun;21(6):536-43. doi: 10.1111/iju.12392. Epub 2014 Feb 16. PMID 24528387
- [Background] Lai HH, Hsu EI, Teh BS, Butler EB, Boone TB. 13 years of experience with artificial urinary sphincter implantation at Baylor College of Medicine. J Urol. 2007 Mar;177(3):1021-5. doi: 10.1016/j.juro.2006.10.062. PMID 17296403
- [Background] John Ware, Jr, Ph.D., Mark Kosinski, M.A., James E. Dewey, Ph.D., Barbara Gandek, M.S. How to score & interpret single item health status measures. Manual for users of SF8, Lincdn, RI. Quality Metric Incorporated, 2001. 1998-2001.
- [Background] Roberts B, Browne J, Ocaka KF, Oyok T, Sondorp E. The reliability and validity of the SF-8 with a conflict-affected population in northern Uganda. Health Qual Life Outcomes. 2008 Dec 2;6:108. doi: 10.1186/1477-7525-6-108. PMID 19055716
- [Background] Moore KN, Jensen L. Testing of the Incontinence Impact Questionnaire (IIQ-7) with men after radical prostatectomy. J Wound Ostomy Continence Nurs. 2000 Nov;27(6):304-12. doi: 10.1067/mjw.2000.110623. PMID 11096410

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03962569/Prot_SAP_000.pdf